CLINICAL TRIAL: NCT04835493
Title: Evaluating Telementoring to Initiate a Multidimensional Diabetes Program for Latino(a)s in Community Clinics: A Randomized Clinical Trial
Brief Title: Evaluating Telementoring for CHW-centered Diabetes Initiatives
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Collaborators: The University of Texas Health Science Center, Houston (Other); University of Houston (Other); Baylor College of Medicine (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 22-0224; R01DK129474 (NIH)
Record Dates: First submitted 2021-04-05; First posted 2021-04-08 (Actual); Last update posted 2025-06-02 (Actual); Status verified 2025-05

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Methods

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: 1. Randomization will be achieved by blinded study staff using an automatic number generator that allows for stratification and blocking.
  2. Individuals entering and obtaining study data will be blinded to study arm
  3. Data will be collected prior to randomization for blinding purposes. Month-12 clinical data will be obtained in-person for both arms by nurses blinded to the study arm e.g., different nurses than those in the group visits, and chart review will be conducted for ADA measurements and for other clinical data if individuals from either study arm do not show.
  4. Blinded research assistants will gather HbA1c, blood pressure, cholesterol, and BMI data for both arms quarterly until 36-months from baseline.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Intervention individuals will receive the 12-month diabetes program
  Interventions: Other: Intervention
- Usual Care (UC) (Other): We will define UC as usual clinical care, which consists of diabetes management provider encounters (mean quarterly) plus monthly individual appointments with a pharm-Ds or nutritionists as clinically indicated. In addition, clinics offer multiple other individual and group opportunities.
  Interventions: Other: Intervention

INTERVENTIONS:
Other: Intervention — In the proposed study, we will conduct a randomized clinical trial of low-income, adult Latino(a)s with type 2 diabetes randomized at the individual level a telehealth-supported, integrated CHWs, medication-access, diabetes education program) (intervention) versus usual care (UC). Our research team will provide telementoring to local clinic teams (providers and CHWs) to initiate the 12-month the program into their clinics.

SUMMARY:
Diabetes care is complex and requires a multidimensional approach, but interventional programs are difficult to initiate in low-income and minority populations. In the proposed study, investigators will mentor local clinics via telehealth to initiate our diabetes program involving telehealth-support, integrated CHWs, medication-access, and diabetes Education into their clinics. Mentoring local clinics to initiate this intervention is a promising strategy to enhance sustainable diabetes care and reduce disparities in vulnerable minority populations.

DETAILED DESCRIPTION:
Diabetes is a major public health problem in Latino(a)s. There are escalating numbers of Latino(a)s diagnosed with diabetes and at disproportionate rates compared to other ethnicities. Numerous interventions have been initiated to improve minority healthcare including diabetes group visits, which have been valuable in improving education and glycemic control. In our group visit investigations, investigators initiated Community Health Workers (CHWs)-local community members who serve as culturally-sensitive patient liaisons to the healthcare system-as part of the multidisciplinary team. Investigators demonstrated that CHWs are vital team members and particularly helpful in identifying medication-access barriers. However, CHWs are frontline workers and often left unsupported and poorly supervised. Investigators used these data to pioneer the combination of four diabetes interventions. This trial showed that individuals randomized to the intervention significantly improved glycemic control, blood pressure and adherence to American Diabetes Association standards compared to usual care. The study also showed that telehealth (mobile health (mHealth) and ZOOM video conferencing) was instrumental in supporting CHWs in their work and enhancing their communication with patients.

The COVID-19 pandemic has highlighted the expansive use of telehealth and its ability to improve healthcare. It has also underscored the pressing need to improve care for low-income minorities. Though diabetes programs are valuable in improving education and clinical outcomes, they are often difficult to initiate in low-income settings. Pragmatic implementation using telehealth to mentor local clinic teams of providers and CHWs is promising to address these barriers. Investigators have pilot data showing the feasibility of telementoring a local clinic to initiate our program that has resulted in improved HbA1c levels but it needs to be tested within a larger sample. In the proposed study investigators will evaluate this approach in a randomized clinical trial (N=320; intervention=160) of low-income, adult Latino(a)s with type 2 diabetes randomized to the diabetes program intervention versus usual care (UC). Our research group will provide telementoring to local clinic teams to initiate our program into their clinics. To evaluate efficacy, investigators will compare the intervention versus UC clinical changes including HbA1c (primary outcome), blood pressure, cholesterol, and body mass index from baseline to 12-months (AIM 1). To compare longitudinal data of study arms, investigators will follow these clinical measures until 36 months (AIM 2). Investigators will also provide program acceptability and evaluation data for participants and clinic teams from baseline to 12-months (AIM 3). Investigators hypothesize that intervention participants will have superior and more sustainable clinical outcomes compared to UC individuals and that the intervention will have high levels of acceptability and evaluation data. Investigators anticipate that the proposed study will provide justification of telementoring to initiate the intervention and strong evidence to improve the longitudinal care of low-income Latino(a)s with diabetes.

ELIGIBILITY:
Inclusion Criteria:

* self-identified Latino(a)
* Spanish-speaking
* >/=18 years
* type 2 diabetes (T2D), e.g., HbA1c >/=6.5%, provider documented T2D, on oral anti-hyperglycemic
* uninsured, <150% federal poverty level

Exclusion Criteria:

* no show to all group visits
* condition that may alter HbA1c levels, e.g., recent blood transfusion
* patients at high-risk or not appropriate for care in a group setting e.g., pregnancy, severe cognitive impairment, frequent clinic appointments for labile glucose/medication titration e.g., insulin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
HbA1c | Baseline to 12-months
  Compare intervention versus control HbA1c levels

SECONDARY OUTCOMES:
Blood pressure | Baseline to 12-months
  Compare intervention versus control blood pressure levels (systolic and diastolic)
Body Mass Index (BMI) | Baseline to 12-months
  Compare intervention versus control BMI levels
Cholesterol | Baseline to 12-months
  Compare intervention versus control cholesterol levels
American Diabetes Association (ADA) adherence measures: Diabetes foot exam | Baseline to 12-months
  Compare intervention versus control adherence to diabetes foot exams
ADA adherence measures: B12 screening | Baseline to 12-months
  Compare intervention versus control adherence to B12 screening
ADA adherence measures: Diabetes eye exam | Baseline to 12-months
  Compare intervention versus control adherence to diabetes eye exams
ADA adherence measures: urine microalbumin screening | Baseline to 12-months
  Compare intervention versus control adherence to urine microalbumin screening
ADA adherence measures: flu vaccination | Baseline to 12-months
  Compare intervention versus control adherence to flu vaccination
ADA adherence measures: statin therapy | Baseline to 12-months
  Compare intervention versus control adherence to statin therapy
Sustainable clinical outcomes: HbA1c | baseline to 36-months
  Compared to control, the intervention will have more sustainable HbA1c levels
Sustainable clinical outcomes: Blood pressure | baseline to 36-months
  Compared to control, the intervention will have more sustainable blood pressure levels (systolic and diastolic)
Sustainable clinical outcomes: BMI | baseline to 36-months
  Compared to control, the intervention will have more sustainable BMI levels
Program satisfaction | 12-months
  Anticipate >/=80% patient satisfaction as demonstrated by our 12-question satisfaction survey questions (on Likert scales of 1 to 10 (n=5 questions) where 10 is very satisfied and 1 is not at all satisfied and from 1-4 (n=3 questions) where 4 is very satisfied and 1 is not satisfied). There are three open-ended questions.
Attrition | baseline to 12-months
  Rate of attrition for intervention participants
Community Health Worker (CHW) knowledge | 12-months
  At 12-months; Knowledge as measured the CHW posttest, which includes 24-questions from the Star Education Study diabetes knowledge test, which has shown validity and reliability in English and Spanish and our TIME 25-question diabetes medication test that has been previously published. Tests are multiple choice with 4 possible answers.
Telehealth Acceptability | 12-months
  Acceptability as measured by the Telehealth Usability Questionnaire, a 21-question survey of telehealth acceptability. Items are ranked on a 5-item scale (1 not acceptable, 5 very acceptable) and divided into six subsections that have shown good to excellent internal consistency.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Vaughan, DO, Principal Investigator — UTMB
Locations (1):
- University of Texas Medical Branch, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No
The NIH policy on data sharing does not apply to this protocol: (1) it is not basic research and involves human subjects, (2) it is anticipated that the data can be readily replicated as the purpose of the study is to train local clinics to conduct the program, (3) more than $500K in direct costs annually are not requested for any year of the protocol.

REFERENCES:
- [Derived] Ameri M, Jabbar LA, Kim S, Raji M, Samson SL, Vaughan EM. Training clinicians to facilitate diabetes group visits. BMC Med Educ. 2025 Feb 25;25(1):309. doi: 10.1186/s12909-025-06876-7. PMID 40001087
- [Derived] Porterfield L, Warren V, Schick V, Gulliot-Wright S, Temple JR, Vaughan EM. Addressing Training Gaps: A Competency-Based, Telehealth Training Initiative for Community Health Workers. Telemed Rep. 2023 Jun 16;4(1):126-134. doi: 10.1089/tmr.2023.0007. eCollection 2023. PMID 37351464

DOCUMENTS (1):
  • Informed Consent Form (2023-06-30): https://cdn.clinicaltrials.gov/large-docs/93/NCT04835493/ICF_000.pdf